CLINICAL TRIAL: NCT03687593
Title: Safety and Performance of Primary Total Knee Arthroplasty Using Legion™ CR Oxinium and CoCr Femoral Implants Combined With Legion™/Genesis™ II XLPE High Flex Tibial Inserts
Brief Title: Safety and Performance Using Legion™ CR Oxinium and CoCr Femoral Implants Combined With Legion™/Genesis™ II XLPE High Flex Tibial Inserts
Acronym: Legion Oxinium
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-4042-10
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Legion™ CR Oxinium and CoCr Femoral Implants combined with Legion™/Genesis™ II XLPE High Flex Tibial Inserts — Single arm study, all subjects received the Legion™ CR Femoral Oxinium and CoCr Implant with Legion™/Genesis™ II XLPE Hi-flex Tibial Insert

SUMMARY:
The purpose of this research is to collect data on patients that had the Legion CR Oxinium and CoCr Femoral Implant and the Legion/Genesis II XLPE High Flex Tibial Inserts implanted in the past. Smith & Nephew will evaluate the safety and performance of these implants.

ELIGIBILITY:
Inclusion Criteria:

1. Subject received primary TKA with the Legion™ CR Femoral Implant (either Oxinium or CoCr) with Legion™/Genesis™ II XLPE Hi-flex Tibial Insert, due to degenerative joint disease (primary diagnosis of osteoarthritis, post-traumatic arthritis, degenerative arthritis, or rheumatoid arthritis).
2. Subject received primary TKA between 24 and 66 months prior to the time of consent.
3. Subject agrees to consent and to follow the study visit schedule (as defined in the study protocol and informed consent form) by signing the IRB/EC approved informed consent form.
4. Subject must be available through ten (10) years postoperative follow-up.

Exclusion Criteria:

1. Subject had Body Mass Index (BMI) > 40 at time of surgery.
2. Subject received the Legion™ CR Femoral Implant with Legion™/Genesis™ II XLPE Hi-flex Tibial Insert as a revision surgery.
3. Subject has a condition that may interfere with the TKA survival or outcome (e.g. Paget's or Charcot's disease, vascular insufficiency, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
4. Subject has a known allergy to one or more of its components of the study device.
5. Subject, in the opinion of the Principal Investigator (PI), has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
6. Subject is entered in another drug, biologic, or device study or has been treated with an investigational product in the past 30 days.
7. Subject is known to be at risk for loss to follow-up, or failure to return for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will screen all subjects who underwent TKA with the LEGION™ CR Oxinium and CoCR Femoral Implants
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Implant survival 10 years postoperatively | 10 years post-op

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Director — Smith & Nephew, Inc.
Locations (4):
- United States (4):
  - Allina Health Systems, Edina, Minnesota
  - ROC Foundation, Reno, Nevada
  - Hawkins Foundation, Greenville, South Carolina
  - Appalachian Orthopedic Associates, Johnson City, Tennessee